CLINICAL TRIAL: NCT04398355
Title: A Clinical Trail of Acupuncture and Liu-Zi-Jue Exercise for Dysphagia in Post-stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Ruijie Ma, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020ZJZS001
Record Dates: First submitted 2020-04-24; First posted 2020-05-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: stroke; dysphagia; rehabilitation; traditional Chinese medicine
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (No Intervention): basic treatment+Swallowing rehabilitation training
- Combination treatment (Experimental): basic treatment+Swallowing rehabilitation training+Chinese traditional rehabilitation
  Interventions: Combination Product: acupuncture; Combination Product: Liu-Zi-Jue Gongfa
- Liu-Zi-Jue treatment (Experimental): basic treatment+Swallowing rehabilitation training+Liu-Zi-Jue
  Interventions: Combination Product: Liu-Zi-Jue Gongfa
- acupuncture treatment (Experimental): basic treatment+Swallowing rehabilitation training+acupuncture
  Interventions: Combination Product: acupuncture

INTERVENTIONS:
Combination Product: acupuncture — acupuncture
  Arms: Combination treatment; acupuncture treatment
Combination Product: Liu-Zi-Jue Gongfa — Liu-Zi-Jue Gongfa
  Arms: Combination treatment; Liu-Zi-Jue treatment

SUMMARY:
The traditional Chinese medicine rehabilitation for post-stroke dysphagia impairment will be intervened, which can promote the recovery of dysphagia function of stroke patients, reduce the disability rate and improve the quality of life.

DETAILED DESCRIPTION:
This study will collect inpatients from April 2020 to December 2022 who from the third affiliated hospital of Zhejiang university of traditional Chinese medicine, Jiaxing hospital of traditional Chinese medicine, Hangzhou hospital of traditional Chinese medicine.this study sets strict time window (stroke recovery, 30-180 days), use multi-center, large sample, randomized controlled study method and the objective recognition rehabilitation evaluation criteria and efficacy evaluation system to evaluate the clinical effect and analysis of health economics.

ELIGIBILITY:
Inclusion Criteria:

* Dysphagia

  * Meet the diagnostic criteria of stroke in traditional Chinese medicine;
  * Meet the diagnostic criteria of ischemic stroke in western medicine;
  * meet the diagnostic criteria of pseudobulbar palsy;
  * Age is 18-85, gender not limited;
  * The course of disease is 30 to 180 days;
  * Water test level 3 and level 3 above;
  * Meet the requirements for indications of acupuncture and moxibustion techniques; Volunteer to participate in this project, the patient has no serious complications, can accept acupuncture treatment and good compliance;
  * Sign informed consent
  * MOCA（Montreal Cognitive Assessment） score above 15.

Exclusion Criteria:

* Dysphagia

  * Patients with true bulbar palsy caused by brainstem encephalitis, motor neurone disease, pontine tumor, multiple sclerosis, myasthenia gravis, medulla bulbar cavity;
  * Cerebral hemorrhage caused by cerebrovascular malformation, trauma, aneurysm and other causes;
  * Pregnant or lactating women;
  * Patients with severe primary chronic diseases, severe dementia and cognitive impairment, serious language understanding disorders, and mental illness, including heart, liver, kidney and other viscera, as well as the endocrine system and hematopoietic system;
  * Suffered from a variety of bleeding tendency diseases;
  * The patient to swallow contrast drug allergy;
  * Patients who do not meet the inclusion criteria, do not have poor treatment compliance as prescribed, cannot judge the efficacy or incomplete data affect the judgment of efficacy and are not suitable for clinical observation;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Swallowing Assessment | Change from Baseline Standardized Swallowing Assessment at 4 weeks
  use Standardized Swallowing Assessment to evaluate the patient's conscious, lip closure control ability, the head and trunk control ability, the respiratory mode.

SECONDARY OUTCOMES:
video fluoroscopic swallowing study score，VFSS score | 0 week；4 weeks
  Mainly includes oral stage, pharynx stage, the degree of pharynx three parts, oral stage for 0-2 points; The pharyngeal period was 0-3 points; The degree of pharynx error is 0-4 points, with a total score of 9 points for the sum of the three points. The higher the score, the better the swallowing function is.
The effective rate of swallowing function treatment | at baseline, 0 week, 4 weeks, 8 weeks and 16 weeks
  The effective rate was calculated according to the score of the standard swallowing function evaluation,scale, and the effective criterion was as follows: the patient's score increased by more than 30% > compared with that before treatment.
Time required for swallowing to improve | at 0 week, 4 weeks, 8 weeks, 16 weeks
  it will be assessed by Water Swallow Test (WST),this test divided into 1 ~ 5 levels. The higher level means less dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: RUIJIE MA, Doctor, Study Director — The Third Affiliated hospital of Zhejiang Chinese Medical University; XINYUN LI, Master, Principal Investigator — Zhejiang Chinese Medical University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Hangzhou hospital of traditional Chinese medicine, Hangzhou, Zhejiang
  - Jiaxing hospital of Chinese traditional medicine, Jiaxing, Zhejiang